CLINICAL TRIAL: NCT01417637
Title: A Randomized Clinical Trial of the Effect of Low Level Laser Therapy in Myofacial Pain Syndrome
Brief Title: The Effect of Low Level Laser Therapy (LLLT) in Myofacial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Dr Farzaneh Ahrari, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88563
Record Dates: First submitted 2011-08-08; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2010-06

CONDITIONS: Myofacial Pain Syndrome
Keywords: TMD; myofacial pain syndrome; low level laser therapy; LLLT
MeSH Terms: conditions — Facial Neuralgia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low level laser (Active Comparator): In this group, the 890 nm diode laser (Ga As) Mustang 2000+, Russia) with frequency of 1500 Hz, and dose of 2 J/cm2 per point in the painful muscles.
  Laser therapy for both the treatment and placebo groups will be applied on all painful muscles three times a week for four weeks.
  Interventions: Radiation: Low level laser therapy
- Placebo (Placebo Comparator): In Group 2 (placebo) the low power laser will be applied with a minimal dose that is very lower than the threshold necessary for therapeutic effects.
  Interventions: Radiation: Placebo group

INTERVENTIONS:
Radiation: Low level laser therapy — Ga As diode laser (890 nm) Mustang 2000+, Russia), with frequency of 1500 Hz, and dose of 2 J/cm2 per point in the painful muscles. Laser therapy will be applied on all painful muscles three times a week for four weeks.
  Other Names: LLLT, myofacial pain syndrome, low power laser
  Arms: low level laser
Radiation: Placebo group — In this group, the low power laser will be applied with a minimal dose that is very lower than the threshold necessary for therapeutic effects. Laser therapy will be applied on all painful muscles three times a week for four weeks.
  Other Names: LLLT, low level laser therapy, myofacial pain
  Arms: Placebo

SUMMARY:
Temporomandibular disorders (TMDs) are the major cause of non-dental pain in orofacial area. Laser therapy can be considered as one of the most recent treatment approaches in the field of physiotherapy. The special features of laser light such as coherence, monochromaticity, and collimation can result in the ability of laser light to modify cellular metabolism, increase tissue repair and reduce edema and inflammation. Several studies demonstrated successful results regarding the use of low level lasers in releasing pain of musculoskeletal conditions, but there are also contradictory reports in this field, and the clinical effectiveness of this treatment modality has been debated in some review articles. A few studies evaluated the efficacy of low level laser therapy in the treatment of temporomandibular disorders and the associated myofacial pain. There are remarkable variations in the methodology of these researches and some reported insufficient data regarding the physical properties of the laser used. The aim of this study is to evaluate the effectiveness of low level laser therapy in improving the sign and symptoms of patients suffering from myofacial pain syndrome.

DETAILED DESCRIPTION:
This study will be implemented on 20 patients referring to Department of Prosthetic Dentistry of Mashhad Dental School. The patients are selected according to the RDC/TMD criteria to include those having temporomandibular disorders with muscular origin. The patients will be randomly assigned to two groups: Group 1 (treatment group) will receive low level laser therapy. The laser light will be applied with 890 nm diode laser (Mustang 2000+, Russia) with frequency of 1500 Hz, and dose of 2 J/cm2 per point in the painful muscles.

In Group 2 (placebo) the low power laser will be applied with a minimal dose that is very lower than the threshold necessary for therapeutic effects. Laser therapy for both the treatment and placebo groups will be applied on all painful muscles three times a week for four weeks. Patients will be evaluated at the start of the treatment, after the 6th and 12th sessions of laser therapy and also one month after the end of the treatment. At each evaluation, the maximum mouth opening with or without pain and masticatory muscle tenderness will be measured. Pain will be measured through the Visual Analogue Scale (VAS). The range of lateral and protrusive mandibular movements, and the difficulty in chewing food will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patients are selected according to the RDC/TMD criteria to include those having temporomandibular disorders with muscular origin.

Exclusion Criteria:

1. Patients with disk displacement (with or without reduction)
2. patients with temporomandibular joint arthralgia or osteoarthritis
3. patients with systemic disease affecting temporomandibular joint
4. patients receiving analgesic or antidepressant drugs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Pain relief | Up to 1 month after laser therapy
  Pain will be measured using visual analogue scale (VAS)

SECONDARY OUTCOMES:
Mouth opening measurement | Up to 1 month after laser therapy
  The maximal mouth opening with and without pain will be measured in mm.
Difficulty of chewing food | Up to 1 month after laser therapy
  A questionare will be used to classify the pain during chewing.

CONTACTS AND LOCATIONS:
Overall Officials: Farzaneh Ahrari, DDS, MS, Principal Investigator — Mashhad University of Medical Sciences
Locations (1):
- Mashhad University of Medical Sciences, Mashhad, Khorasan, Iran